CLINICAL TRIAL: NCT00168870
Title: Randomized Phase II Study to Compare a Combination Therapy With Gemcitabine and Treosulfan Versus a Monotherapy as First-Line Chemotherapy for Patients With Metastatic Ocular Melanoma
Brief Title: Study of Metastatic Ocular Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Haema CBF AHM UK/AS 04
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2007-08-31 (Estimated); Status verified 2006-09

CONDITIONS: Ocular Melanoma
Keywords: metastatic ocular melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Gemcitabine; treosulfan

INTERVENTIONS:
Drug: Gemcitabine
Drug: Treosulfan

SUMMARY:
This study evaluates treatment with combination versus monotherapy for patients with metastatic ocular melanoma.

DETAILED DESCRIPTION:
Treatment of patients with metastatic ocular melanoma with combination chemotherapy Gemcitabine and Treosulfan versus monotherapy with Treosulfan as first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic ocular melanoma

Exclusion Criteria:

* Prior treatment with chemotherapy
* Active 2nd malignancy
* Cerebral metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2003-02

PRIMARY OUTCOMES:
Determination of efficacy according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria

SECONDARY OUTCOMES:
Time to progression

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Keilholz, MD, Principal Investigator — Charité Campus Benjamin Franklin Berlin
Locations (1):
- Hematology & Oncology Charité CBF Berlin, Berlin, State of Berlin, Germany